CLINICAL TRIAL: NCT02939365
Title: Precision Medicine Offers Belatacept Monotherapy (PROBE)
Brief Title: Precision Medicine Offers Belatacept Monotherapy
Acronym: PROBE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Because of inability to get FDA approval for
Sponsor: University of California, San Francisco (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Flavio Vincenti, Professor of Clinical Medicine, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM103-382
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Transplantation
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belatacept patients (Experimental): Forty patients who are previously enrolled in belatacept based regimens with a minimum of 7 years of follow up at 4 transplant centers and who are maintained on belatacept, an antiproliferative ± steroids will be approached for enrollment.
  Drug withdrawal of steroids (in patients on steroids) and of antiproliferatives (MPAs or mTor inhibitors). Patients who continue to be stable for 3 months on belatacept monotherapy will be converted from q 4 weeks to q 8 weeks belatacept administrations.
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Belatacept — The transition to belatacept monotherapy and possibly to q 8 weeks administration can be safely done by applying personalized (i.e. precision) medicine. This includes phenotypic analysis of lymphocyte subsets, a quiescent molecular profiling of blood and urine prior to drug withdrawal and immune monitoring with KSORT after stepwise withdrawal of steroids and antiproliferatives. Furthermore, trough PK of belatacept will be measured for conversion to q 8 week therapy for discovering research purposes.
  Other Names: Nulojix®

SUMMARY:
The purpose of this study is to determine the safety and feasibility of converting patients to Belatacept monotherapy (receiving just one immunosuppression drug), and to see what percentage of those patients can be safely converted to once every 8 week administration of Belatacept. Belatacept has been approved by the Food and Drug Administration (FDA) for kidney transplant recipients.

DETAILED DESCRIPTION:
Patients on belatacept who fulfill the entry criteria will be screened to determine if they have a quiescent molecular immunologic profile with kSORT and uCRM. Patients who screen negative on all 2 tests will undergo stepwise withdrawal first of steroids then of MMF or mTor inhibitors. Prior to each withdrawal the 2 screening molecular tests will be performed and advancement to the next withdrawal phase will be performed if both are negative. Patients who are maintained on belatacept monotherapy with quiescent kSORT and uCRM and elevated kSPOT will be transitioned to q 8 weeks belatacept administration.

Forty patients who are previously enrolled in belatacept based regimens with a minimum of 7 years of follow up at 4 transplant centers and who are maintained on belatacept, an antiproliferative ± steroids will be approached for enrollment.

Drug withdrawal of steroids (in patients on steroids) and of antiproliferatives (MPAs or mTor inhibitors) will follow the design shown in the Study Schema. Patients who continue to be stable for 3 months on belatacept monotherapy will be converted from q 4 weeks to q 8 weeks belatacept administrations.

ELIGIBILITY:
Inclusion Criteria:

* Stable renal function with a GFR ≥ 35 ml/min
* No history of acute rejection
* A spot urine protein creatinine ratio of 0.5 or less
* No DSA

Entry: Biomarker criteria

* Blood kSORT and urine CRM tests that are quiescent at entry and following each drug withdrawal.
* A third biomarker KSPOT will be used to assess if any patients has achieved tolerance.

Eligibility for 8 week Belatacept Administration

* Trough levels of belatacept at 4 weeks of greater than 2 µg/ml
* Trough levels of belatacept at 8 weeks of equal or greater than 1 µg/ml

Exclusion Criteria:

* Patients with < eGFR (35 ml/min)
* History of rejection
* Protein/creatinine rate >0.5
* Presence of DSA

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Percent patients converted to belatacept | 12 months
  To determine the percent of patients that can be safely converted to belatacept monotherapy
Percent patients safely converted to q8 week administration | 12 months
  2. To determine the percent of patients on belatacept monotherapy that can be safely converted to 8 week administration of belatacept

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Vincenti, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No